CLINICAL TRIAL: NCT01611441
Title: Investigation of Biomarkers in an Exploratory Study in Patients With Osteoarthritis of the Knee Undergoing Total Knee Replacement Surgery
Brief Title: Investigation of Specific Protein/Markers in Patients With Osteoarthritis of the Knee Having a Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2285M00029; D2285M00029
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis of the knee; Biomarkers
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, urine, synovial fluid, synovial membrane, cartilage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with osteoarthritis of the knee: Patients with osteoarthritis of the knee undergoing total knee replacement surgery.

SUMMARY:
The main purpose of the study is to better understand how specific proteins/markers in blood, urine, synovial fluid (a lubricating fluid secreted by the membrane lining the joints), and joint tissue are involved in osteoarthritis of the knee. The aim is to investigate if there is a correlation between x-ray results, specific proteins/markers and different types of pain in patients with osteoarthritis of the knee. The study consists of 3 visits over 3-20 days and the last visit will be the day of surgery.

DETAILED DESCRIPTION:
Investigation of Biomarkers in an Exploratory Study in Patients with Osteoarthritis of the Knee Undergoing Total Knee Replacement Surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo a total knee replacement due to osteoarthritis.
* Symptoms of the knee for at least 6 months prior to study start.

Exclusion Criteria:

* Key-hole surgery performed on target knee within 3 months prior to study start.
* History of disorders in which part of the immune system is missing or defective.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary and secondary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with upregulation of IL-6 or the IL-6 signalling pathway in the knee. | 3-20 days prior to day 1 (surgery) and day 1 (surgery) .

SECONDARY OUTCOMES:
Biomarkers in synovial fluid, synovial membrane, and cartilage. | Day 1 (surgery).
Biomarkers in blood and urine. | 3-20 days prior to day 1 (surgery) and day 1 (surgery).
Biomarkers by Magnetic Resonance Imaging (MRI). | 1-5 days prior to day 1 (surgery).
Polymorphisms in 10 specific genes. | 3-20 days prior to day 1 (surgery) or at any time in the study.
WOMAC (Western Ontario and McMaster Osteoarthritis Index) variables and NPQ (Neuropathic Pain Questionnaire) variables. | 3-20 days prior to day 1 (surgery) and 1-5 days prior to day 1 (surgery).
  WOMAC consists of 3 subscales with a total of 24 questions regarding pain, stiffness and difficulty in performing daily activities. A VAS (Visual Analogue Scale) will be used for the patient to report the severity of the symptoms on the target knee. Endpoints are marked "No pain" (0 mm) and " Extreme pain" (100 mm) on a paper PRO (Patient Reported Outcome) questionnaire. The less pain scored the better outcome.
  NPQ accesses 12 different pain intensities. 0 represents no intensity and 100 represents worst intensity imaginable. The less intensity the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, MD, PHD, Study Director — AstraZeneca R&D Sodertalje, Sweden
Locations (6):
- Canada (3):
  - Research Site, Montreal
  - Research Center, Newmarket
  - Research Site, Québec
- Sweden (3):
  - Research Site, Kungälv
  - Research Site, Motala
  - Research Site, Stockholm

REFERENCES:
- [Derived] Radojcic MR, Thudium CS, Henriksen K, Tan K, Karlsten R, Dudley A, Chessell I, Karsdal MA, Bay-Jensen AC, Crema MD, Guermazi A. Biomarker of extracellular matrix remodelling C1M and proinflammatory cytokine interleukin 6 are related to synovitis and pain in end-stage knee osteoarthritis patients. Pain. 2017 Jul;158(7):1254-1263. doi: 10.1097/j.pain.0000000000000908. PMID 28333699